CLINICAL TRIAL: NCT06322771
Title: Women's Refusal to Participate in a Randomized Trial Involving First-trimester Screening for Pre-eclampsia: Factors Associated With Refusal and Reasons for Acceptance and Refusal
Acronym: RANSPRE-refus
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240376
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related
Keywords: Refusal; Clinical trial; Factors; Reasons; Pregnancy; Pre-eclampsia
MeSH Terms: conditions — Treatment Refusal; Pre-Eclampsia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Refusal: A questionnaire will be given to patients who have refused to participate in the RANSPRE trial
  Interventions: Behavioral: Questionnaire
- Acceptance: A questionnaire will be given to patients who have agreed to participate in the RANSPRE trial
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire about acceptance
  Groups: Acceptance
Behavioral: Questionnaire — Questionnaire about refusal
  Groups: Refusal

SUMMARY:
The main objective is to assess whether there are factors associated with women's refusal to participate in a randomized clinical trial involving first-trimester screening for pre-eclampsia. The secondary objective is to qualitatively evaluate the reasons for acceptance and refusal to participate.

DETAILED DESCRIPTION:
1. Determine the acceptance/refusal rate among all women identified, eligible and offered RCT.
2. Comparison of demographic characteristics between the two groups

   * Group 1: women accepting to participate in RCT
   * Group 2: women refusing to participate in RCT
3. Assessment of motivations for acceptance (based on questionnaire given to women who agree to participate)
4. Evaluation of reasons for refusal to participate - obstacles (based on the questionnaire given to women who refuse to participate).

ELIGIBILITY:
Inclusion Criteria :

Inclusion criteria are the same as for the RANSPRE trial.

Any pregnant woman is eligible if:

* monofetal pregnancy
* between 11 and 14 weeks
* legal age
* health insurance coverage

Exclusion Criteria :

Inclusion criteria are the same as for the RANSPRE trial. A history of pre-eclampsia in a previous pregnancy and a contraindication to aspirin are non-inclusion criteria.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women identified and eligible to participate in the RANSPRE trial within the Port-Royal maternity ward and having their T1 ultrasound scan within the maternity ward will be included.
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Factors associated with women's refusal | Day 1
  The primary objective is to assess whether there are factors associated with women's refusal to participate in the RANSPRE randomized clinical trial.

SECONDARY OUTCOMES:
Number of acceptations | Day 1
Number of refusals | Day 1
Demographic characteristics | Day 1
Questionnaire "acceptance" | Day 1
  Evaluation of motivations linked to acceptance (based on the questionnaire given to women who agree to participate)
  The secondary objective is to qualitatively assess the reasons for acceptance of participation.
Questionnaire "refusal" | Day 1
  Evaluation of the reasons for refusing to participate - obstacles (based on the questionnaire given to women who refuse to participate).
  The secondary objective is to qualitatively assess the reasons for refusal of participation.

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Athiel, MD, Principal Investigator — Port-Royal Maternity - APHP
Locations (1):
- Port-Royal Maternity, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No